CLINICAL TRIAL: NCT00956423
Title: Exercise: A Novel Treatment for Obstructive Sleep Apnea
Brief Title: Comparison of Physical Activity Regimens as Treatments for Obstructive Sleep Apnea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Christopher Kline, PI, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R36CD000695-01 (NIH)
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; exercise training; aerobic exercise; resistance exercise
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- moderate-intensity exercise training (Experimental)
  Interventions: Behavioral: moderate-intensity aerobic and resistance training
- low-intensity stretching (Active Comparator)
  Interventions: Behavioral: low-intensity stretching

INTERVENTIONS:
Behavioral: moderate-intensity aerobic and resistance training — Individuals will complete four days of aerobic exercise of moderate intensity (60% of maximal VO2, approximated from heart rate). Duration of aerobic activity will gradually increase from weeks 1 through 4 until 180 min of aerobic exercise at the prescribed intensity is performed each week. Following aerobic exercise on two days per week, moderate-intensity resistance training will be performed using eight different resistance machines. One set of 8-12 repetitions will be performed during weeks 1-4; from week 5-on, 2 sets of 8-12 repetitions will be performed.
  Arms: moderate-intensity exercise training
Behavioral: low-intensity stretching — Individuals will perform supervised whole-body flexibility exercises on two days per week. Two sets of each exercise will be performed, with the duration of each stretch gradually increasing from 15 sec to 30 sec. A total of 15-20 stretches, focusing on whole-body flexibility, will be performed.
  Arms: low-intensity stretching

SUMMARY:
The purpose of this study is to compare the efficacy of two different physical activity regimens as complementary or alternative treatment options for the treatment of obstructive sleep apnea. A secondary purpose of the study is to examine the effects of these activity regimens on various health consequences of obstructive sleep apnea, including blood pressure, systemic inflammation, and daytime functioning.

ELIGIBILITY:
Inclusion Criteria:

* moderate-intensity obstructive sleep apnea (AHI >= 15)
* sedentary status

Exclusion Criteria:

* current treatment for obstructive sleep apnea (CPAP, oral devices, etc.)
* significant cardiovascular, pulmonary, or metabolic disease
* uncontrolled hypertension
* inability to exercise (e.g., musculoskeletal, neuromuscular, orthopedic problems)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Laboratory polysomnographic assessment of apnea-hypopnea index | pre- and post-intervention (12 weeks later)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Kline, MS, Principal Investigator — University of South Carolina, William Jennings Bryan Dorn VA Medical Center; Shawn D Youngstedt, PhD, Study Chair — University of South Carolina, William Jennings Bryan Dorn VA Medical Center
Locations (2):
- United States (2):
  - University of South Carolina, Columbia, South Carolina
  - William Jennings Bryan Dorn VA Medical Center, Columbia, South Carolina

REFERENCES:
- [Background] Norman JF, Von Essen SG, Fuchs RH, McElligott M. Exercise training effect on obstructive sleep apnea syndrome. Sleep Res Online. 2000;3(3):121-9. PMID 11382910
- [Background] Giebelhaus V, Strohl KP, Lormes W, Lehmann M, Netzer N. Physical Exercise as an Adjunct Therapy in Sleep Apnea-An Open Trial. Sleep Breath. 2000;4(4):173-176. doi: 10.1007/s11325-000-0173-z. PMID 11894204
- [Background] Ueno LM, Drager LF, Rodrigues AC, Rondon MU, Braga AM, Mathias W Jr, Krieger EM, Barretto AC, Middlekauff HR, Lorenzi-Filho G, Negrao CE. Effects of exercise training in patients with chronic heart failure and sleep apnea. Sleep. 2009 May;32(5):637-47. doi: 10.1093/sleep/32.5.637. PMID 19480231
- [Background] Quan SF, O'Connor GT, Quan JS, Redline S, Resnick HE, Shahar E, Siscovick D, Sherrill DL. Association of physical activity with sleep-disordered breathing. Sleep Breath. 2007 Sep;11(3):149-57. doi: 10.1007/s11325-006-0095-5. PMID 17221274
- [Background] Peppard PE, Young T. Exercise and sleep-disordered breathing: an association independent of body habitus. Sleep. 2004 May 1;27(3):480-4. doi: 10.1093/sleep/27.3.480. PMID 15164902
- [Derived] Kline CE, Ewing GB, Burch JB, Blair SN, Durstine JL, Davis JM, Youngstedt SD. Exercise training improves selected aspects of daytime functioning in adults with obstructive sleep apnea. J Clin Sleep Med. 2012 Aug 15;8(4):357-65. doi: 10.5664/jcsm.2022. PMID 22893765
- [Derived] Kline CE, Crowley EP, Ewing GB, Burch JB, Blair SN, Durstine JL, Davis JM, Youngstedt SD. Blunted heart rate recovery is improved following exercise training in overweight adults with obstructive sleep apnea. Int J Cardiol. 2013 Aug 20;167(4):1610-5. doi: 10.1016/j.ijcard.2012.04.108. Epub 2012 May 8. PMID 22572632
- [Derived] Kline CE, Crowley EP, Ewing GB, Burch JB, Blair SN, Durstine JL, Davis JM, Youngstedt SD. The effect of exercise training on obstructive sleep apnea and sleep quality: a randomized controlled trial. Sleep. 2011 Dec 1;34(12):1631-40. doi: 10.5665/sleep.1422. PMID 22131599